CLINICAL TRIAL: NCT01154894
Title: Double-blind Randomized Placebo-controlled Trail
Brief Title: Dietary Fatty Acids Improve Social Impairment in Autism Spectrum Disorders
Acronym: Fatty acid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ashiya University (Other)
Responsible Party: Kunio Yui, Ashiya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KunioYui
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2008-12

CONDITIONS: Autism Spectrum Disorders
Keywords: arachidonic acid; autism spectrum disorders; social interaction; randomized controlled trial; DHA
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo-controlled trial (Experimental)
  Interventions: Other: Aravita including arachidonic acid and docosaheaenoic acid

INTERVENTIONS:
Other: Aravita including arachidonic acid and docosaheaenoic acid — Nine of 13 Participants were treated with 6 capsules of Aravita per day for 16-week trial, remaining 4 participants aged under 12 years received 3 capsules per day.

SUMMARY:
In a double-blind, placebo-controlled 16-week trial investigators administered daily doses of either youths with autism spectrum disorders.ARA and DHA supplementation significantly improved communication as well as social withdrawal symptoms. This pilot study provides the first evidence that supplementation with larger ARA doses added to DHA improve impaired social interaction in youths with Autism Spectrum Disorders (ASD).

DETAILED DESCRIPTION:
We recruited 13 individuals who met the DSM-IV criteria for a diagnosis of high functioning autistic disorder (n=1) or Asperger's Disorder (n=12),corroborated by the Autism Diagnostic Interview-Revised. Participants were free of any medical or comorbid psychiatric disorders. Other inclusion criteria included weigh of at least 16 kg, either a verbal or performance intelligence quotient (IQ) above 80, and a score greater than 10 on the social withdrawal subscale of the Aberrant Behavior Checklist-Community.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of high functioning autistic disorder or Asperger's Disorder. Free of any medical or comorbid psychiatric disorders.

Exclusion Criteria:

* Any medical treatment for other psychiatric disorders

Ages: 6 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-community (ABC) | Pretreatment and at 4 weeks after intervention for 16-weeks trial
  ABC is used to estimate abnormal behavior, including 5 subscales, irritability, social withdrawal, stereotypy, hyperactivity, and inappropriate speech

SECONDARY OUTCOMES:
Social Responsiveness Scale (SRS) | pretreatment and at 4 weeks after intervention for 16-weeks trial
  The SRS is assessed the severity of social communication impairment in any population.

REFERENCES:
- [Derived] Yui K, Koshiba M, Nakamura S, Kobayashi Y. Effects of large doses of arachidonic acid added to docosahexaenoic acid on social impairment in individuals with autism spectrum disorders: a double-blind, placebo-controlled, randomized trial. J Clin Psychopharmacol. 2012 Apr;32(2):200-6. doi: 10.1097/JCP.0b013e3182485791. PMID 22370992